CLINICAL TRIAL: NCT07361029
Title: Phase Ia Study of a LentiGen® CD19 Chimeric Antigen Receptor (CAR) T Cells in Adult Patients With Relapsed/Refractory CD19 Positive Acute Lymphoblastic Leukemia (ALL) Using a Closed Transduction System
Brief Title: CD19 Chimeric Antigen Receptor (CAR) T Cells in Adults With Relapsed/Refractory CD19 Positive Acute Lymphoblastic Leukemia
Acronym: CD19 CART CELL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Principal Investigator, Riad El Fakih, Consultant, Lymphoma / Myeloma, King Faisal Specialist Hospital & Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2191207
Record Dates: First submitted 2025-08-27; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Relapsed Refractory Acute Lymphoblastic Leukemia
Keywords: CD19 CAR T; relapsed/refractory acute lymphoblastic leukemia (ALL).
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Chimeric Antigen Receptor (CAR)-modified T cell (CD19)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm dose finding (Experimental)
  Interventions: Other: CAR T cells chimeric antigen receptor cells

INTERVENTIONS:
Other: CAR T cells chimeric antigen receptor cells — CAR T Cells

SUMMARY:
This is a Phase Ia, open label, dose finding single center trial designed to evaluate the maximum tolerated dose, safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of CD19 CAR T cells targeting the B cell surface antigen CD19 following administration of chemotherapy lymphodepletion regimen in adults (age 18 - 75) with relapsed/refractory acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
Approximately 24 patients are planned to be enrolled in four cohorts during the dose-escalation stage. Within each cohort, 3 patients will receive treatment with CD19 CAR T cells.

The starting dose level is 5x10*5cells/kg, administered as a single dose by IV infusion. Dose escalation will proceed in accordance with the dose-escalation Dose-escalation decisions will be made by the Data Safety Monitoring Board (DSMB) in consultation with the investigators . CD19 CAR T cells administration between the first and second patient in each dose level will be separated by a minimum of 4 weeks. CD19 CAR T cells administration between each subsequent patient in a dose level will be separated by a minimum of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 to 75 years old (patients is older than 18.0 and less than 75.0 years old) 2. Signed informed consent form 3. Ability to comply with the study protocol 4. Relapsed/refractory B-cell acute lymphoblastic leukemia (B-ALL):

  1. Second or greater bone marrow (BM) relapse; or
  2. Primary refractory, defined as not achieving complete remission (CR) after 2 cycles of a standard chemotherapy regimen, or Chemo-refractory, defined as not achieving CR after 1 cycle of standard chemotherapy for relapsed leukemia; or
  3. Philadelphia chromosome-positive ALL intolerant of or with 2 failed lines of tyrosine kinase inhibitor (TKI) therapy; or
  4. Relapsed patients ineligible for Allogeneic Stem Cell Transplant (AlloSCT) due to lack of a suitable donor.
  5. Relapsed after AlloSCT. at least 12 weeks after alloSCT or relapse happened after withdrawing the post-transplant immunosuppression
  6. Relapsed after prior CAR T cell and still CD19 positive. . (Patients with a history of ≥grade CRS, ≥ grade 3 ICANS, or severe hypersensitivity reactions following prior CAR T-cell therapy should be excluded.) 5. BM with ≥5% lymphoblasts by morphologic assessment at screening 6. For relapsed patients, documentation of CD19 tumor expression in BM or peripheral blood by flow cytometry or immunohistochemistry within 1 month of study entry 7. Patients with a history of CNS or meningeal involvement must be in a documented clinical remission prior to registration.

     8. Alanine aminotransferase (ALT) ≤5 times the upper limit of normal for age 9. Bilirubin ≤2 x ULN 10. Patients with good renal function defined as Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 cc/min.

     11. Absolute Neutrophil Count (ANC): Patients must have an ANC ≥ 1.0 x 109

     /L without the use of growth factors 12. Platelet Count: Patients must have a platelet count ≥ 50 x 109/L without transfusion support within 7 days of screening.

     13. Absolute Lymphocyte Count: Patients must have an absolute lymphocyte count ≥ 0.5 x 109/L.

     14. Definition of Adequate Organ Function:
     * Renal Function: Glomerular Filtration Rate (GFR) > 60mL/min.
     * Hepatic Function: AST/ALT ≤ 5 x ULN and bilirubin ≤ 2 x ULN. Total bilirubin 1.5 ULN (except Gilbert's syndrome).
     * Pulmonary Function: Adequate respiratory function defined as oxygen saturation ≥ 93% on room air.
     * Cardiac Function: Left ventricular ejection fraction (LVEF) ≥ 45% by echocardiogram or MUGA scan and QTcF ≤ 480 ms. 15. Minimum level of pulmonary reserve defined as grade ≤1 dyspnea and pulse oxygenation >93% on room air 16. Left ventricular ejection fraction ≥45% confirmed by echocardiogram within 30 days of screening 17. Karnofsky ≥ 70% and /or ECOG 0-2 at the time of screening 18. Women of child bearing age should have negative serum pregnancy test within 7 days prior to enrollment 19. If sexually active:

  <!-- -->

  1. Females should use effective birth control 1 month prior to screening until 12 months after CAR T cell infusion
  2. Males to use condom for six months after infusion 20. Meet institutional criteria to undergo leukapheresis or have an acceptable, stored leukapheresis product

Exclusion Criteria:

1. Clinically Active central nervous system (CNS) involvement by malignancy
2. History or presence of uncontrolled underlying seizure disorder not related to B-ALL
3. History of or active clinically significant cardiovascular dysfunction, including any of the following:

   * History of stroke within 24 months prior to the CD19 CAR T cells infusion or with ongoing sequelae
   * History of transient ischemic attack within 12 months prior to the CD19 CAR T cells infusion
   * History of myocardial infarction within 36 months prior to the CD19 CAR T cells infusion
   * Symptomatic congestive heart failure (NYHA class III/IV), unstable angina pectoris, cardiac arrhythmia requiring therapy
   * Uncontrolled arrhythmias, or history of or active ventricular arrhythmia requiring medication
   * Active or history of coronary heart disease that remains symptomatic
   * Active or history of unstable or stable angina
   * Left ventricular ejection fraction (LVEF) < 45% confirmed by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA) scan
4. Creatinine clearance < 60
5. Concomitant genetic syndromes associated with Bone Marrow (BM) failure states, such as Fanconi anemia, Kostmann syndrome, Schwachman syndrome, or any other BM failure syndrome; patients with Down syndrome are not excluded
6. Burkitt lymphoma/leukemia
7. Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and no evidence of active disease
8. Treatment with any prior gene therapy product (except prior CAR-T cell therapy)
9. Positive HIV test within 8 weeks of screening
10. Serologic status reflecting active hepatitis B or C infection: Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded.)
11. Received an investigational medicinal product on trial within the 30 days prior to screening
12. Pregnant
13. Lactating
14. Women of child-bearing potential and all male participants, unless using highly effective methods of contraception for 1 year after CAR-T infusion
15. Therapeutic systemic doses of steroids (>=0.5mg/kg prednisone equivalent) must be stopped >72 hours prior to lymphodepletion
16. TKIs and hydroxyurea must be stopped >72 hours prior to lymphodepletion
17. The following drugs must be stopped >1 week prior to lymphodepleting chemotherapy:

    vincristine, 6- mercaptopurine, 6-thioguanine, methotrexate 2 weeks prior to CART infusion: salvage chemotherapy (e.g., clofarabine, cytosine arabinoside >100 mg/m2

    , anthracyclines, cyclophosphamide, methotrexate ≥25 mg/m2

    ), excluding the required lymphodepleting chemotherapy drugs
18. Pegylated asparaginase must be stopped >4 weeks prior to CAR T cell infusion
19. CNS disease prophylaxis and/or intrathecal chemotherapy must be stopped >1 week prior to CAR T cell infusion
20. Radiation therapy at non-CNS site must be completed >2 weeks prior to CAR T Cell infusion
21. CNS-directed radiation must be completed >8 weeks prior to CAR T cell infusion
22. Known History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study (including, but not limited to, cyclophosphamide and fludarabine used in the lymphodepleting chemotherapy, DMSO used as a cryoprotectant in the cell media, etc.)
23. Autologous transplant within 6 weeks of planned CAR-T cell infusion
24. Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy.
25. Primary Immunodeficiency Patients:

    • Patients with known primary immunodeficiency disorders are excluded due to increased risk of adverse outcomes.
26. Recent Live Vaccine Administration:

    * Patients who have received a live vaccine within 4 weeks prior to enrolment are excluded.
    * Additionally, vaccination with live vaccines is not recommended for at least 6 weeks prior to the start of lymphodepleting chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | throughout study completion, Day1 to 5 years
  To assess the maximum tolerated dose, safety and tolerability of intravenous infusion of CD19 CAR T cells using based on incidence, nature, and severity of AEs graded according to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5 (NCI CTCAE v5), cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS).

SECONDARY OUTCOMES:
Evaluate the success rate of product manufacturing | Pre-infusion
  To evaluate the success rate of product manufacturing based on product meeting release criteria
preliminary anti-tumor activity of CD19 CAR T cells in treated patients | Day30 and Day 60
  Preliminary anti-tumor activity of CD19 CAR T post-infusion and Minimal residual disease (MRD) status at 1st-month and 2nd- month post-infusion in treated patient
Safety of CD19 CAR T cells | Day 1- 8, Day 14-21, Day30, Day60, Day90, Day120, Day180, Day270, and yearly
  Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.
Safety of CD19 CAR T cells | Day 1- 8, Day 14-21, Day30, Day60, Day90, Day120, Day180, Day270, and yearly]
  Number of Participants with Treatment Related immune effector cell-associated neurotoxicity syndrome (ICANS). will be graded according to ASTCT criteria.
safety of CD19 CAR T cells | Day 1- 8, Day 14-21, Day30, Day60, Day90, Day120, Day180, Day270, and yearly
  Number of Participants with Treatment-Related cytokine release syndrome (CRS)
To characterize the pharmacokinetic (PK) profile of CD19 CAR T cells | Day7, Day14, Day28, 2month, 4 month, 6month,10month,12month 14month,16month,18month,20month, 22month, and 24month
  To characterize the pharmacokinetic (PK) profile of CD19 CAR T cells using area under the curve (AUC)
To characterize the pharmacokinetic (PK) profile of CD19 CAR T cells | Day7, Day14, Day28, 2month, 4 month, 6month,10month,12month 14month,16month,18month,20month, 22month, and 24month
  To characterize the pharmacokinetic (PK) profile of CD19 CAR T cells using maximum concentration (Cmax)
To characterize the pharmacokinetic (PK) profile of CD19 CAR T cells | Day7, Day14, Day28, 2month, 4 month, 6month,10month,12month 14month,16month,18month,20month, 22month, and 24month
  To characterize the pharmacokinetic (PK) profile of CD19 CAR T cells using minimum concentration (Cmin)
To characterize the pharmacokinetic (PK) profile of CD19 CAR T cells | Day7, Day14, Day28, 2month, 4 month, 6month,10month,12month 14month,16month,18month,20month, 22month, and 24month
  To characterize the pharmacokinetic (PK) profile of CD19 CAR T cells using clearance (Cl)
To characterize the pharmacokinetic (PK) profile of CD19 CAR T cells | Day7, Day14, Day28, 2month, 4 month, 6month,10month,12month 14month,16month,18month,20month, 22month, and 24month
  To characterize the pharmacokinetic (PK) profile of CD19 CAR T cells using volume (V)
To characterize the pharmacokinetic (PK) profile of CD19 CAR T cells | Day7, Day14, Day28, 2month, 4 month, 6month,10month,12month 14month,16month,18month,20month, 22month, and 24month
  To characterize the pharmacokinetic (PK) profile of CD19 CAR T cells using half-life (T1/2)

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital and Research Center, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
yes with Miltenyi our collaborator